CLINICAL TRIAL: NCT05754281
Title: The PRECISION II Study: Evaluating the Accuracy of the LabPatch Glucose Sensing System in Insulin-treated Patients With Diabetes
Brief Title: The PRECISION II Study: Evaluating the Accuracy of the LabPatch Glucose Sensing System
Status: Recruiting | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Cambridge Medical Technologies, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00000130
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: LabPatch Continuous Glucose Monitoring (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: 60 adult subjects with type 1 or type 2 diabetes treated with insulin. The accuracy of the 2nd Gen LabPatch Continuous Glucose Sensing will be evaluated during the study visit, comparing to YSI 2300 STAT Plus, OneTouch Verio and FreeStyle Lite.
  Interventions: Device: 2nd Gen LabPatch Glucose Sensing System

INTERVENTIONS:
Device: 2nd Gen LabPatch Glucose Sensing System — I. The 2nd Gen LabPatch chip which lies in the center of a clasp unit. The chip measures approximately 15.7 mm [0.618"] x 15.7 mm [0.618"]. The chip has a telescopic micropipette which draws interstitial fluid to be analyzed for glucose levels. The chip is also able to measure skin temperature to ensure appropriate skin contact
  II. A LabPatch clasp device
  III. A wire that connects the clasp unit to a Windows tablet which will communicate with the clasp via an application. Each data point will be viewed on the tablet and the application will also have some limited graphing capabilities to view trends of previous measurements

SUMMARY:
The purpose of this study is to evaluate the accuracy of the Cambridge Medical Technologies, LLC second generation (2nd Gen) LabPatch glucose sensing system compared to a laboratory glucose analyzer (YSI 2300 STAT Plus) and 2 commercial glucometers, OneTouch Verio and Freestyle Lite. The primary endpoint of this study is the mean absolute relative difference (MARD) for 2nd Gen LabPatch system compared to each of the above mentioned glucose references over a 6 hour outpatient visit.

DETAILED DESCRIPTION:
In a pilot study conducted previously by our group using the prototype 1st generation LabPatch system (PRECISION study, 2016-31), the investigators found that LabPatch glucose measurements strongly correlated with those of YSI, OneTouch Verio, and Freestyle lite in a sample of 30 subjects. However, the investigators observed significant inter- and intra-subject variability of LabPatch glucose measurements. Factors that may have contributed to this variability include: manual manufacturing of the 1st Gen LabPatch circuit chips and/or variability in the pressure applied by subjects on the circuit chip at each measurement. To control for these variables with the goal of improving overall accuracy, Cambridge Medical Technologies, LLC significantly improved and completely automated the manufacturing process of the circuit chips. In addition, the system has been miniaturized to a more user-friendly layout and with a clasp unit to control for pressure applied by the subject finger on the circuit chip.

The 2nd Gen LabPatch system consists of:

I. The 2nd Gen LabPatch chip which lies in the center of a clasp unit. The chip measures approximately 15.7 mm [0.618"] x 15.7 mm [0.618"]. The chip has a telescopic micropipette which draws interstitial fluid to be analyzed for glucose levels. The chip is also able to measure skin temperature to ensure appropriate skin contact II. A LabPatch clasp device III. A wire that connects the clasp unit to a Windows tablet which will communicate with the clasp via an application. Each data point will be viewed on the tablet and the application will also have some limited graphing capabilities to view trends of previous measurements The system has been previously tested on 10 human subjects with type 1 diabetes, each for six hours, at the Georgetown University Medical Center under clinical conditions supervised by a medical team including an endocrinologist and dermatologist. The test confirmed the absence of pain or abnormal physical sensation and that the operation of the device causes no tissue damage,instigates no neural sensation for the subject, and leaves no blemish on the skin. No skin damage incurred by the LabPatch operation was detected.

The 2nd Gen LabPatch system is an in vitro diagnostic device (IVD), does not have significant risk and is therefore exempted from the IDE requirements. In addition, the device uses an in vitro diagnostic technology that does not create adverse events and therefore a data safety monitoring board (DSMB) is not requited.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.
2. Subject is between 18 and 75 years of age.
3. Subject is diagnosed with type 1 diabetes or type 2 diabetes for ≥3 months and is being treated with insulin injections in the form of multiple daily injections or through insulin infusion pump.
4. Subject is a male or a non-pregnant and non-lactating female, at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to screening visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

1. Subject is pregnant or lactating.
2. Subject is not treated with insulin.
3. Subject has/had acute or chronic, contagious, infectious disease
4. Subjects with history of blood-born chronic viral infection (e.g. Hepatitis C and HIV)
5. Subject has/had clotting or bleeding disorders or other hematological disease.
6. Subject has an active malignancy (excluding the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in-situ of the cervix).
7. Subject had a recent cardiovascular event (e.g., myocardial infarction, stroke) ≤ six months prior to screening visit; or stated history of congestive heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with type 1 or type 2 diabetes treated with insulin.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean absolute relative difference (MARD) | Baseline, every 15 minutes for a total of 6 hours
  Blood glucose values (mg/dL) from the LabPatch system and reference YSI, One Touch Verio, and FreeStyle Lite will be used to report the mean absolute relative difference (MARD) in Percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No